CLINICAL TRIAL: NCT03635411
Title: Basis: Evaluating Sirtuin Supplements To Benefit Elderly Trauma Patients
Brief Title: Basis: Evaluating Sirtuin Supplements To Benefit Elderly Trauma Patients (BES2T BET)
Acronym: BestBet
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elysium Health (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 829947
Record Dates: First submitted 2018-08-07; First posted 2018-08-17 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Recovery of Function
MeSH Terms: interventions — nicotinamide-beta-riboside; Pterocarpus marsupium; Radial Basis Function Networks

STUDY DESIGN:
Intervention Model Description: Assessing Safety and Tolerability
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basis (Experimental): Nicotinamide riboside 500 mg and pterostilbene 100 mg given twice daily in divided doses for 90 days
  Interventions: Dietary Supplement: Nicotinamide Riboside and Pterostilbene
- Placebo (Placebo Comparator): Placebo given twice daily for 90 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside and Pterostilbene — Nicotinamide riboside and pterostilbene manufactured by Basis
  Other Names: Basis; NRPT
  Arms: Basis
Dietary Supplement: Placebo — Sugar pill manufactured to mimic Basis supplement.
  Arms: Placebo

SUMMARY:
Basis: Evaluating Sirtuin Supplements To Benefit Elderly Trauma Patients (BES2T BET) A phase I, randomized, double-blind, placebo-controlled, single institutional pilot trial investigating the impact of nicotinamide riboside/pterstilbene (BasisTM) on functional recovery after traumatic fall in elderly patients

.

DETAILED DESCRIPTION:
This Phase I pilot study will determine if supplementing with the combination of NR and Pter (BasisTM) is well tolerated and will provide the pretrial data necessary to plan a randomized clinical trial aimed at determining if BasisTM improves the functional outcome of injured elderly patients.

Primary Objective

• To determine if BasisTM is well tolerated by elderly patients up to 90 days post injury

Secondary Objectives:

* To determine if BasisTM preserves or improves muscular strength, endurance, and activity following traumatic injury in elders.
* To determine if BasisTM preserves or improves physiologic composition (muscle/fat ratio) following traumatic injury in elders.
* To determine if BasisTM decreases 90 day incidence of recurrent falls
* To determine the impact of BasisTM on subjective well-being (pain) and quality of life (EQ-5D-5L)
* To determine if BasisTM alters NAD and sirtuin activity in inflammatory cells.

Elderly trauma patients who present after a traumatic injury will be screened and enrolled within 48 hours of their trauma evaluation. Baseline status will be determined using functional surveys, physical assessments, and physiologic measurements. Patients will be randomized to either BasisTM or placebo for 90 days. Patients will be reassessed at 2 weeks, 6 weeks (optional) and 90 days. Activity and heart rate will be monitored continuously using a wrist FitBit Device.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 65 year old
2. Patient presenting to trauma bay

Exclusion Criteria:

1. Currently taking medication for severe to moderate dementia (see Appendix 9)
2. Currently taking niacin, nicotinic acid, nicotinamide, or nicotinamide riboside
3. Pre-existing immobility (wheel chair or bed bound)
4. Renal failure requiring hemodialysis or peritoneal dialysis
5. End-stage Liver Disease (Model for End Stage Liver Disease Score ≥ 25) (see Appendix 11)
6. Intubated prior to enrollment (excluding intubation for surgery)
7. More than 48 hours post-injury
8. Thoracic Anatomic Injury Score > 3 (see Appendix 10)
9. Other Injuries with Anatomic Injury Score >2, excluding thorax (see Appendix 10)
10. Hip fractures
11. Non-English speaking

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-12-06 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Complications | 90 days
  To analyze patient complications through daily adverse event monitoring and summarize adverse events for each arm

SECONDARY OUTCOMES:
Grip Strength Scores | 90 days
  To measure if BasisTM preserves or improves grip strength using Jamar hand dynamo-meter in non-dominant hand
Inhalation Volume Measurements | 90 days
  To measure if BasisTM preserves or improves lung volume by measuring inhaled volumes using incentive spirometry
6 Minute Timed Walk Test Scores | 90 days
  To measure if BasisTM preserves or improves 6 minute Timed Walk Test according to the AmericanThoracic Society Guidelines.
Timed Get Up and Go Test Scores | 90 days
  To measure if BasisTM preserves or improves timed get up and go scores
Measurement of Muscle/ Fat Ratio | 90 days
  To measure if BasisTM preserves or improves physiologic composition (muscle/fat) ratio) using bioelectric impedance
Incidence of Adverse Events | 90 days
  To analyze if BasisTM decreases 90 day incidence of recurrent falls
Incidence of Pain and Daily Pain Medication Dosage | 90 days
  To analyze the impact of BasisTM on subjective well-being pain through measurement of pain medication amounts and frequency.
Analysis of Quality of Life Scores | 90 days
  To analyze the impact of BasisTM on subjective well-being through analysis of EuroQol 5 Dimensions-5 Levels (EQ-5D-5L) scores and EuroQol Visual Analogue Scale (EQ Vas). EQ-5D-5L Scores consist of 5 sections: Mobility, Self-Care, Usual Activities, Pain/ discomfort and Anxiety/ Depression. The minimum score in each is 1, and the maximum is 5, where 5 indicates extreme problems and 1 indicates no problems. A total of 3125 possible health states exist and each stats is referred to in terms of a 5 digit code. State 11111 indicates no problems on any of the 5 dimensions, whereas state 12345 indicates no problems with mobility, slight problems with washing or dressing, moderate problems with doing usual activities, severe pain or discomfort and extreme anxiety or depression. The EQ-VAS is scored from 0 to 100 where 0 means the worst health you can imagine and 100 means the best health you can imagine.
Late Life Function and Disability Instrument Scores analysis as a measure of subject independence, function, and disability | 90 days
  To analyze the impact of BasisTM on subjective well-being through analysis of Late Life Function and Disability Scores. Questions are scored on a scale of 5 to 1, where 1 means no difficulties with function and 1 means patients are unable to complete the functions on their own. Disability questions are scored from 1 to 5, where 1 means subjects do not complete activities and feel limited and 5 means subjects can complete activities and don't feel at all limited. Scores are computed using the LLFDI Scoring Software.
Analysis of scores on Mini Mental Status Exam as a measure of cognitive function and dementia | 90 days
  To analyze the impact of BasisTM on subjective well-being through analysis of Mini Mental Status Scores. The maximum score is 30 and the sections are orientation (10 points), registration (3 points), attention and calculation (5 points), recall (3 points), language and praxis (9 points). 0 is the lowest and 30 is the best score.
Analysis of subject nutrition through Mini Nutritional Assessment Scores | 90 days
  To analyze the impact of BasisTM on subjective well-being through analysis of Mini Nutritional Assessment scores. The maximum score is 14 points and the lowest (worst score) is 0.
Analysis of Subject independence using Barthel Index scores | 90 days
  To analyze the impact of BasisTM on subjective well-being through analysis of Barthel Index Scores. The index consists of 10 Activities of daily living, 8 of which represent activities related to personal care while 2 are related to mobility. The index yields a total score out of 100 with higher scores indicating greater degrees of functional independence.
Analysis of patient comorbidities as a measure of adverse events in evaluating Basis tolerability | 90 days
  To analyze the impact of BasisTM on subjective well-being through analysis of Charlson comorbidity index scores. The CCI accounts for 19 pre-defined comorbid conditions and is given a different weight depending on each's association with 1-year mortality. The total score in CCI is determined by the combined weight of the patient's conditions, where higher scores represent worse conditions.
Analysis of inflammatory cell activity | 90 days
  To measure if BasisTM alters Nicotinamide adenine dinucleotide (NAD) and sirtuin activity in inflammatory cells. Liquid chromatography mass spectrometry will assay for NAD.
Analysis of Mitochondrial Function | 90 days
  Mitochondrial content will be determined by citrate synthase activity. Mitochondrial respiration and the generation of reactive oxygen species will be measured using high-resolution respirometry and fluoremtry.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Sims, Principal Investigator — Univeristy of Pennsylvania
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No